CLINICAL TRIAL: NCT02816320
Title: Validity of Information Employed to Generate Standardized Mortality Ratios Using Hospital Administrative Databases (RNMH)
Acronym: RNMH
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL15_0175
Record Dates: First submitted 2016-06-22; First posted 2016-06-28 (Estimated); Last update posted 2019-04-03 (Actual); Status verified 2019-04

CONDITIONS: Surgical Condition; Obstetrical Condition; Hospitalization in Acute Care
Keywords: hospital mortality; standardized mortality ratios; patient safety; healthcare quality; hospital performance; administrative data
MeSH Terms: interventions — Hospitalization

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Inpatient stays: All patients who were hospitalized in participating hospitals in France during the study period were eligible for inclusion.
  Interventions: Other: Hospitalization

INTERVENTIONS:
Other: Hospitalization — Patients who were hospitalized in acute care

SUMMARY:
In a retrospective cross-sectional study, investigators aimed to valid the variables employed to generate standardized mortality ratio from hospital administrative databases. For this purpose, investigators have compared those variables collected in administrative databases with the information available in patient medical record.

ELIGIBILITY:
Inclusion Criteria:

* All inpatients stays in acute care from high mortality diagnosis related groups (DRGs) registered in administrative databases of participating hospitals from January to December 2010.

Exclusion Criteria:

* Hospital participation refusal

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: A random sample of patients who were hospitalized in 24 participating hospitals during the study period.
Sampling Method: Probability Sample
Enrollment: 715 (Actual)
Dates: Start 2014-07; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
In-hospital mortality | within 90 days of admission (D90)
  Death collected in hospital administrative databases at the end of in patient stay